CLINICAL TRIAL: NCT04736160
Title: Pilot Study: hCG Secreted by Blastocyst as Potential Marker of Embryo Quality
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: IVI Vigo (Other)
Collaborators: Instituto Valenciano de Infertilidad, IVI VALENCIA (Other)
Responsible Party: Sponsor
Other Study IDs: 1709-VGO-092-EM
Record Dates: First submitted 2021-01-29; First posted 2021-02-03 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-01

CONDITIONS: Embryo Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: collect data — The data for this project will be obtained directly from the IVI digital work platform (SIVIS) where the characteristics and scans performed to each patient are recorded. Furthermore, it will be recollected information from the time-lapse incubator. For the current study will be used Embryoscope and Geri time-lapse incubators

SUMMARY:
hCG is a hormone produced very early by the pre-embryo, but not by the oocyte. It has a pivotal role in the trophoblast differentiation, and embryo implantation as well as the corpus luteum support. In spite of its well-known role, the literature about it is scarce.

The aim of this study is to evaluate the relation between the amount of hCG secreted by the blastocyst and embryo euploidy status and morphological pre-embryo quality according to morphokinetic pattern.

We will analyse the amount of hCG secreted by blastocyst to the culture medium thorough mass spectrometry and it will be correlated with the main morphokinetic issues and the chromosomal structure after NGS analysis at blastocyst stage.

We will take the pre-embryo spent culture medium that has been discarded after embryo culture without any interference on the pre-embryo neither any different deviation of standard protocol of embryo manipulation. Furthermore, the evaluation by time-lapse technology will let to document the main issues of embryo development, also without any deviation of the standard protocol.

We are waiting to find the value of hCG secreted by blastocyst as a potential marker of embryo quality and ploidy status.

DETAILED DESCRIPTION:
Embryo selection based on morphological and morphokinetic characteristics seems to be insufficient to guarantee implantation. For this reason, in recent years, it has appeared new embryo selection strategies to increase the success of assisted reproduction treatments.

Human chorionic gonadotrophin (hCG) is a glycoprotein hormone composed of two subunits, alpha and beta, non-covalently attached. It is secreted by the blastocyst trophoblastic cells and because it is detectable in maternal blood shortly after embryo implantation and it can be used as a pregnancy marker (Cole et al., 1987).

Historically, it has been believed that the only function of hCG was to stimulate the secretion of progesterone by the corpus luteum. Nowadays, we know that it also plays a key role in the invasion, fusion of the endometrium by the blastocyst and the angiogenesis. In addition, it has a paracrine role to induce trophoblast differentiation (Cole, 2009).

Recently, it has been proposed that its concentration would be linked to the time after implantation and to the number of trophoblastic cells (Tanbo and Eskild, 2015). However, the concentration of hCG shows considerable variations among embryos, and it has been postulated that this could be due to differences in the implantation potential at the second week of embryo development (Lopata and Oliva, 1993). Then, hCG could be a good marker in embryo selection. In fact, it is already known that there is a higher secretion of hCG by those blastocysts that present more adherence to the culture plate compare with those that do not present it (Dokras et al., 1991).

In addition, this hormone presents variants that change as the blastocyst grows. The early embryos secreted more acidic variants than the more advanced ones (Lopata, 1997), and it has recently been shown that the different isoforms correspond to different degrees of glycosylation and metabolic degradation. The measurement of the concentration of these isoforms can be indicate to predict embryo implantation (Butler et al., 2013).

Despite all this, there are few studies published that measure the concentration of hCG in the culture medium and most of them are published more than 15 years ago (Hay and Lopata, 1988; Lopata and Hay, 1989; Dokras et al., 1991; Lopata and Oliva 1993). This fact, together with the need to optimize the embryo classification, makes us consider whether it could be a good candidate as an embryo/aneuploidy selection marker.

ELIGIBILITY:
Inclusion criteria:

* Age < 42.
* BMI < 30kg/m2.
* SET (Single embryo transfer)

Exclusion Criteria:

* Hydrosalpinx.
* Any indication of oocyte vitrification

Ages: 18 Years to 41 Years | Sex: Female
Age Groups: Adult
Study Population: Patients undergoing IVF with indication of PGT-A and time-lapse evaluation
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2018-12-05 (Actual); Primary Completion 2019-11-25 (Actual); Study Completion 2021-11-25 (Estimated)

PRIMARY OUTCOMES:
To evaluate the relation between the amount of hCG secreted by blastocyst and morphological embryo quality according to morphokinetic pattern. | Since 2018 to april 2020
  hCG secreted by blastocyst as a potential marker of embryo quality and ploidy status.

CONTACTS AND LOCATIONS:
Overall Officials: Elkin Muñoz, Study Director — IVI Vigo
Locations (1):
- IVI Vigo, Vigo, Pontevedra, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Basile N, Vime P, Florensa M, Aparicio Ruiz B, Garcia Velasco JA, Remohi J, Meseguer M. The use of morphokinetics as a predictor of implantation: a multicentric study to define and validate an algorithm for embryo selection. Hum Reprod. 2015 Feb;30(2):276-83. doi: 10.1093/humrep/deu331. Epub 2014 Dec 19. PMID 25527613
- [Background] Dominguez F, Gadea B, Esteban FJ, Horcajadas JA, Pellicer A, Simon C. Comparative protein-profile analysis of implanted versus non-implanted human blastocysts. Hum Reprod. 2008 Sep;23(9):1993-2000. doi: 10.1093/humrep/den205. Epub 2008 Jun 12. PMID 18556682
- [Background] Meseguer M, Herrero J, Tejera A, Hilligsoe KM, Ramsing NB, Remohi J. The use of morphokinetics as a predictor of embryo implantation. Hum Reprod. 2011 Oct;26(10):2658-71. doi: 10.1093/humrep/der256. Epub 2011 Aug 9. PMID 21828117